CLINICAL TRIAL: NCT00702780
Title: Multi-center, Randomized, Placebo-controlled, Double-blind Clinical Trial of Escitalopram on the Progression Delaying Effect in Alzheimer's Disease
Brief Title: Progression Delaying Effect of Escitalopram in Alzheimer's Disease
Acronym: ESAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Dong Young Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUDC001
Record Dates: First submitted 2008-06-15; First posted 2008-06-20 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; escitalopram; MRI
MeSH Terms: conditions — Alzheimer Disease | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Experimental): Escitalopram 20mg tablet by mouth once a day
  Interventions: Drug: escitalopram
- Placebo (Placebo Comparator): Placebo 20mg tablet by mouth once a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: escitalopram — 5 mg/day for 2 weeks, 10 mg/day for 2 weeks and 20 mg/day for 48 weeks (maintaining donepezil at the previous stable dose during the whole trial period)
  Other Names: Lexapro
  Arms: Escitalopram
Drug: placebo — 5mg/day for 2 weeks, 10mg/day for 2 weeks and 20mg/day for 48 weeks (maintaining donepezil at the previous stable dose during the whole trial period)
  Arms: Placebo

SUMMARY:
This study aimed to test whether escitalopram would slow the brain atrophy in patients with mild to moderate AD over the 52-week period.

DETAILED DESCRIPTION:
* Study institutions: Four university hospitals in Korea
* Design: Multi-center, randomized, placebo-controlled, double-blind clinical trial
* Subjects: 74 probable Alzheimer's disease patients who have been taking donepezil at stable dose within 2 months (Escitalopram 37 : Placebo 37)

ELIGIBILITY:
Inclusion Criteria:

* Age:40~90 years
* Education:not illiterate
* Clinical Dementia Rating (CDR):0.5~2
* Modified Hachinski Ischemic Score (Rosen et al., 1979):less than 4
* Dementia according to DSM-IV criteria
* Probable Alzheimer's disease according to NINCDS-ADRDA criteria
* Current ongoing donepezil medication at stable doses (5 ~ 10 mg/day) for at least 2 months

Exclusion criteria:

* Evidence of delirium, confusion or altered consciousness
* Evidence of Parkinson's disease, stroke, brain tumor and normal pressure hydrocephalus
* Evidence of infectious or inflammatory brain disease
* Evidence of serious cerebrovascular diseases
* Current major depressive disorder or other major psychiatric illnesses
* Evidence of serious or unstable medical illnesses which can significantly change cognitive state
* History of alcohol or other substance dependence
* Any antidepressant medications within the previous 4 weeks
* Absence of a reliable and cooperative collateral informant
* Any conditions which prohibit MRI scan, such as presence of pacemaker or cerebrovascular clip, and claustrophobia
* Evidence of focal brain lesions on MRI including lacunes and white matter hyperintensity lesions of grade 2 or more by Fazeka scale

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Young Lee, MD, PhD, Principal Investigator — Dept. of Neuropsychiatry, Seoul National University Hospital & Seoul National University College of Medicine; Jong Inn Woo, MD, PhD, Principal Investigator — Dept. of Neuropsychiatry, Seoul National University Hospital & Seoul National University College of Medicine
Locations (4):
- South Korea (4):
  - Kangwon National University Hospital, Chuncheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Konkuk University Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Escitalopram: escitalopram 20mg qd
- Placebo: placebo 20mg qd
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 37 | 37
Completed | 28 | 29
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.33 (7.12) | 74.82 (9.19) | 74.58 (8.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: % Change of Hippocampus Volume
Time Frame: 52 weeks
Population: The analysis was performed for per-protocol (PP) population, which included participants who had both baseline and follow-up MRI scan suitable for analysis.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 28 | 29
percentage of change | -7.63 (7.32) | -7.28 (5.76)

2. Primary Outcome: % Change of Whole Brain Volume
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 28 | 29
percentage of change | -3.27 (2.69) | -2.30 (3.08)

ADVERSE EVENTS:
Time Frame: Baseline, and 2, 4, 8, 16, 28, 40, 52 weeks after baseline.
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 2/37 | 3/37
Other Adverse Events (participants affected / at risk) | 13/37 | 7/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=37) | Placebo (N=37)
Jaundice (Hepatobiliary disorders) | 1 | 0
Death by traffic accident (Social circumstances) | 1 | 0
Cerebral hemorrhage (Vascular disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=37) | Placebo (N=37)
dizziness (Nervous system disorders) | 4 | 0
vomiting (Gastrointestinal disorders) | 0 | 1
anorexia (Gastrointestinal disorders) | 1 | 1
abdominal pain (Gastrointestinal disorders) | 0 | 1
diarrhea (Gastrointestinal disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
somnolence (General disorders) | 1 | 0
tremor (Nervous system disorders) | 1 | 0
fall (Injury, poisoning and procedural complications) | 0 | 1
violent behavior (Psychiatric disorders) | 1 | 0
urinary incontinence (Renal and urinary disorders) | 1 | 0
hypoglycemia (Endocrine disorders) | 1 | 0
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No